CLINICAL TRIAL: NCT05136300
Title: Pulmonary Rehabilitation After Minimal Invasive Surgery in Lung Cancer
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Lars Dinjens, MD, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABR 63724
Record Dates: First submitted 2021-11-17; First posted 2021-11-29 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Lung Cancer; Surgery
MeSH Terms: conditions — Lung Neoplasms | interventions — Pain Clinics

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An integrated multidisciplinary rehabilitation program on general quality of life (short form 36, SF-36, subdomain general health) in the 12 months postoperative period in patients undergoing elective minimal invasive surgery in lung cancer
  Interventions: Behavioral: Pulmonary rehabilitation
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — Patients in the intervention group will receive physical therapy, scheduled pain monitoring and coaching by a social worker.
  The intensity of the rehabilitation training program will be determined separately for each patient by a steepramp and 1-repetition test within 3 weeks post-operative. The intervention group will be trained and educated in 2 sessions of 2 hours per week, for a period of 3 months.
  Other Names: Pain clinic
  Arms: Intervention

SUMMARY:
Morbidity in the post-operative phase of pulmonary surgery is characterised by impairment due to pain, dyspnoea and loss of exercise tolerance. We demonstrated previously that rehabilitation after thoracotomy is limited due to pain. Since minimal invasive surgery is the new standard in lung cancer, resulting in a reduction of postoperative pain, we believe there are new possibilities for post-operative integrated multidisciplinary rehabilitation in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective, minimal invasive surgery with intention to cure.
2. Age between 18 and 80 years.
3. ECOG 0 - 2 post-surgery.

Exclusion Criteria:

1. Patients with chronic pain
2. Previous pulmonary surgery
3. Comorbidity limiting rehabilitation

   1. Rheumatoid arthritis
   2. Severe ischaemic heart disease or myocardial failure; EF ≤ 35 %.
   3. Muscle disease
   4. Fibromyalgia
   5. Neurologic disorders (Parkinson disease, CVA and lesions of the spinal cord)
   6. Psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (SF-36) | 12 months
  effects of an integrated multidisciplinary rehabilitation program on general quality of life

SECONDARY OUTCOMES:
SGRQ | 12 months
  health-related quality of life
VAS | 12 months
  post-operative pain
WHO-PS | 12 months
  performance score
6 minute walking distance | 12 months
  exercise tolerance
international physical activity questionnaire, iPAQ | 12 months
  physical activity

CONTACTS AND LOCATIONS:
Overall Officials: J Stigt, Principal Investigator — Isala
Locations (1):
- Isala, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: No